CLINICAL TRIAL: NCT05637970
Title: A Prospective Randomized Study Comparing the Time to Ambulation (TTA) and Safety of Using a Closure Device Alone and in Conjunction With a Potassium Ferrate Pad (StatSeal Advanced) Following Transcatheter Aortic Valve Replacement (TAVR) Via the Transfemoral Artery
Brief Title: Comparing Perclose to Statseal With Perclose in Transcatheter Aortic Valve Replacement Arteriotomy Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Olcay Aksoy, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-000961
Record Dates: First submitted 2022-11-23; First posted 2022-12-06 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Arterial Occlusion; Cardiovascular Diseases; Hematoma
MeSH Terms: conditions — Arterial Occlusive Diseases; Cardiovascular Diseases; Hematoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Perclose Only (Active Comparator): Patients will have a PercloseTM device deployed at the arteriotomy. Manual pressure will be held for at least five minute, the beginning of which will correspond to time point zero. Patent hemostasis will be documented after device deployment. Any manual compression needed or per protocol under the disgression of the operator will count towards the time to hemostasis. After hemostasis is achieved in the cath lab the patient will be sent to the post-operative area for monitoring. If any additional bleeding is appreciated, manual compression will again be held. If any new bleeding from the puncture site or under the skin the patient will again lay supine and at least 10 minutes of manual pressure will be held. This will be continued until the patient has no bleeding.
  Interventions: Device: Perclose
- Perclose with Statseal Device (Experimental): Patients will have a PercloseTM device deployed at the arteriotomy. A Statseal disc will applied and manual pressure will be held for at least five minute, the beginning of which will correspond to time point zero. Patent hemostasis will be documented after device deployment. Any manual compression needed or per protocol under the disgression of the operator will count towards the time to hemostasis. After hemostasis is achieved in the cath lab the patient will be sent to the post-operative area for monitoring. If any additional bleeding is appreciated, manual compression will again be held. If any new bleeding from the puncture site or under the skin the patient will again lay supine and at least 10 minutes of manual pressure will be held. This will be continued until the patient has no bleeding.
  Interventions: Device: Perclose; Device: Statseal

INTERVENTIONS:
Device: Perclose — Patients will have a PercloseTM device deployed at the arteriotomy. Manual pressure will be held for at least five minute, the beginning of which will correspond to time point zero. Patent hemostasis will be documented after device deployment. Any manual compression needed or per protocol under the disgression of the operator will count towards the time to hemostasis. After hemostasis is achieved in the cath lab the patient will be sent to the post-operative area for monitoring. If any additional bleeding is appreciated, manual compression will again be held. If any new bleeding from the puncture site or under the skin the patient will again lay supine and at least 10 minutes of manual pressure will be held. This will be continued until the patient has no bleeding.
  Other Names: Suture based hemostasis device
Device: Statseal — Patients will have a PercloseTM device deployed at the arteriotomy. A Statseal disc will applied and manualpressure will be held for at least five minute, the beginning of which will correspond to time point zero. Patent hemostasis will be documented after device deployment. Any manual compression needed or per protocol under the disgression of the operator will count towards the time to hemostasis. After hemostasis is achieved in the cath lab the patient will be sent to the post-operative area for monitoring. If any additional bleeding is appreciated, manual compression will again be held. If any new bleeding from the puncture site or under the skin the patient will again lay supine and at least 10 minutes of manual pressure will be held. This will be continued until the patient has no bleeding.
  Other Names: potassium ferrate disc with topical hydrophilic polymer
  Arms: Perclose with Statseal Device

SUMMARY:
The purpose of this clinical study is to compare how well two different devices achieve hemostasis in patients undergoing a transfemoral transcatheter aortic valve replacement. Both devices are approved by the FDA for this use, and have already been used by clinicians on patients undergoing transfemoral procedures. It is believed that the use of both devices in combination compared to the Perclose alone will shorten the time that it takes to 'seal' the artery, resulting in a shorter period of time that manual pressure will be held, shorter procedure time and less complications after the procedure.

ELIGIBILITY:
Inclusion Criteria:

Delivery of a 14-16 French Transcatheter aortic valve replacement system

Exclusion Criteria:

* Use of a hemostasis method or device besides PercloseTM (Perclose may not be used in situations of heavy calcification, presence of dissection, etc).
* Use of an anticoagulant other than unfractionated heparin or bivalirudin during the procedure.
* Any use of glycoprotein inhibitors or cangrelor.
* Use of sheathless guides.
* Any anticipated need for continued anticoagulation post-catheterization, including extended bivalirudin infusion.
* Any active treatment with oral anticoagulants continued during course of procedure.
* Presence of arteriovenous dialysis fistula in the ipsilateral leg.
* Any physical deformity or trauma / injury of the leg that would prevent proper placement or function of the hemostasis band.
* Inability of the patient to personally consent for the study. (no surrogate consent)
* Cardiogenic shock, emergent procedures (high risk myocardial infarctions), or any clinical instability as assessed by the physician performing the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Ronald Reagan Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Perclose Only: Patients will have a PercloseTM device deployed at the arteriotomy. Manual pressure will be held for at least five minute, the beginning of which will correspond to time point zero. Patent hemostasis will be documented after device deployment. Any manual compression needed or per protocol under the disgression of the operator will count towards the time to hemostasis. After hemostasis is achieved in the cath lab the patient will be sent to the post-operative area for monitoring. If any additional bleeding is appreciated, manual compression will again be held. If any new bleeding from the puncture site or under the skin the patient will again lay supine and at least 10 minutes of manual pressure will be held. This will be continued until the patient has no bleeding.
  Perclose: Patients will have a PercloseTM device deployed at the arteriotomy. Manual pressure will be held for at least five minute, the beginning of which will correspond to time point zero. Patent hemostasis will be documented after device deployment. Any manual compression needed or per protocol under the disgression of the operator will count towards the time to hemostasis. After hemostasis is achieved in the cath lab the patient will be sent to the post-operative area for monitoring. If any additional bleeding is appreciated, manual compression will again be held.
Period: Overall Study
Arm/Group | Perclose Only | Perclose With Statseal Device
Started | 26 | 24
Completed | 26 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Perclose Only: Patients will have a PercloseTM device deployed at the arteriotomy. Manual pressure will be held for at least five minute, the beginning of which will correspond to time point zero. Patent hemostasis will be documented after device deployment. Any manual compression needed or per protocol under the disgression of the operator will count towards the time to hemostasis. After hemostasis is achieved in the cath lab the patient will be sent to the post-operative area for monitoring. If any additional bleeding is appreciated, manual compression will again be held. If any new bleeding from the puncture site or under the skin the patient will again lay supine and at least 10 minutes of manual pressure will be held. This will be continued until the patient has no bleeding.
  Perclose: Patients will have a PercloseTM device deployed at the arteriotomy. Manual pressure will be held for at least five minute, the beginning of which will correspond to time point zero. Patent hemostasis will be documented after device deployment. Any manual compression needed or per protocol under the disgression of the operator will count towards the time to hemostasis. After hemostasis is achieved in the cath lab the patient will be sent to the post-operative area for monitoring.
- Total: Total of all reporting groups
Arm/Group | Perclose Only | Perclose With Statseal Device | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.2 (6.8) | 80.0 (7.3) | 79.6 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 17 | 16 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis
Description: From the time of manual compression after PercloseTM deployed until hemostasis is achieved without complication.
Time Frame: 24 hours post procedure (± 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Perclose Only | Perclose With Statseal Device
Number analyzed (Participants) | 26 | 24
minutes | 5.11 (4.4) | 4.3 (4.4)

2. Secondary Outcome: Patients With Hematoma
Description: Presence of small <5cm, medium 5-10cm, or large >10cm hematoma based on physical exam or diagnostic imaging.
Time Frame: 24 hours post procedure (± 1 hour)
Measure: Count of Participants; unit: Participants
Arm/Group | Perclose Only | Perclose With Statseal Device
Number analyzed (Participants) | 26 | 24
Participants
  Small <5cm | 0 | 0
  Medium 5-10cm | 0 | 0
  Large >10cm | 1 | 1

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Perclose Only | Perclose With Statseal Device
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT05637970/Prot_SAP_002.pdf